CLINICAL TRIAL: NCT04590781
Title: A Phase 1b/2 Multiple-Dose Study to Evaluate the Safety and Efficacy of XmAb18087 ± Pembrolizumab in Subjects With Advanced Merkel Cell Carcinoma or Extensive-stage Small Cell Lung Cancer (DUET-1-02) Protocol
Brief Title: Safety and Efficacy of XmAb18087 ± Pembrolizumab in Advanced Merkel Cell Carcinoma or Extensive-stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study has been terminated early by the sponsor due to business decision.
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb18087-02; DUET 1-02 (Other: Xencor)
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Merkel Cell Carcinoma; Small Cell Lung Cancer
Keywords: MCC; SCLC
MeSH Terms: conditions — Carcinoma, Merkel Cell; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: XmAb18087 Monotherapy (Experimental): Part A, will enroll participants with previously treated advanced MCC, consists of safety-run in cohorts followed by an expansion cohort.
  Interventions: Biological: XmAb18087
- Part B: XmAb18087 + pembrolizumab (Experimental): Part B, will enroll participants with advanced MCC not previously treated with anti-programmed cell death 1 (PD1) or anti-programmed cell death ligand 1 (PDL1) agents, consists of safety run-in cohorts followed by an expansion cohort.
  Interventions: Drug: XmAb18087 ± Pembrolizumab
- Part C: XmAb18087 monotherapy (Experimental): Part C will enroll participants with previously treated extensive-stage SCLC and consists of safety-run in cohorts followed by an expansion cohort.
  Interventions: Biological: XmAb18087

INTERVENTIONS:
Biological: XmAb18087 — Monoclonal bispecific antibody
  Arms: Part A: XmAb18087 Monotherapy; Part C: XmAb18087 monotherapy
Drug: XmAb18087 ± Pembrolizumab — XmAb18087 ± Pembrolizumab
  Arms: Part B: XmAb18087 + pembrolizumab

SUMMARY:
This is a Phase 1b/2, multiple-dose study designed to describe safety and efficacy, and to assess PK and immunogenicity of XmAb18087 monotherapy and in combination with pembrolizumab in participants with metastatic Merkel cell (MCC) or locoregional MCC that has recurred after locoregional therapy with surgery and/or radiation therapy, and mAb18087 monotherapy in participants with extensive-stage small cell lung cancer (SCLC) that has progressed after standard therapies.

This study was terminated by the sponsor. No participants enrolled in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Adult participants ≥ 18 years
* Disease measurable by RECIST 1.1 criteria using either computed tomography (CT) or magnetic resonance imaging (MRI) scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* All participants must have adequate archival tumor sample (slides or archival formalin-fixed paraffin-embedded [FFPE] block[s] containing tumor that has not been previously irradiated
* Female participants of childbearing potential must agree to use a highly effective method of birth control during and for 4 weeks after completion of study. success), or sexual abstinence
* Fertile male participants must be willing to practice a highly effective method of birth control for the duration of the study and continuing for 4 weeks after the last dose of XmAb18087 or pembrolizumab (when applicable
* Able and willing to complete the entire study according to the study schedule

Additional Inclusion Criteria for Part A and Part B Cohorts:

• Histologically or cytologically confirmed metastatic MCC or locoregional MCC that has recurred following standard locoregional therapy with surgery and/or radiation therapy.

Additional Inclusion Criteria for Part A Cohorts:

• Participants must have progressed on or been ineligible for treatment with anti-PD1 or anti-PDL1 therapy.

Additional Inclusion Criteria for Part B Cohorts:

• Participants must be eligible to receive pembrolizumab as standard of care.

Additional Inclusion Criteria for Part C Cohorts:

• Histologically or cytologically confirmed extensive-stage SCLC that has progressed following standard therapies

Exclusion Criteria:

Additional Exclusion Criteria for Part B Cohorts: XmAb18087 in Combination with Pembrolizumab

* Prior treatment with therapeutics directed at anti-programmed cell death 1 (anti-PD1) or anti-programmed cell death ligand 1 (anti-PDL1)
* Have severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Thompson, MD, PhD, Study Director — Medical Director, Clinical Development, Xencor
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering, New York, New York
  - OU Health, Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been terminated early by the sponsor. No participants with advanced Merkel Cell Carcinoma (MCC) not previously treated with anti-programmed cell death 1 (PD1) or anti-programmed cell death ligand 1 (PDL1) agents were enrolled for Part B.
Groups:
- Part A: XmAb18087 Monotherapy: Participants with previously treated advanced MCC were administered XmAb18087 Monotherapy.
- Part C: XmAb18087 Monotherapy: Participants with previously treated extensive-stage SCLC were administered XmAb18087 monotherapy.
Period: Overall Study
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of XmAb18087.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: No data is reported here to maintain participant confidentiality.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: No data is reported here to maintain participant confidentiality.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: A treatment-emergent adverse event (TEAE) was any untoward medical occurrence in a participant treated with study drug. The TEAE does not necessarily have a causal relationship with this treatment. A TEAE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. TEAEs may include the onset of new illness and the exacerbation of preexisting conditions. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section."
Time Frame: Day 1 (after dosing) up to end of study (up to 163 days)
Population: All participants who received at least 1 dose of XmAb18087. No participants were enrolled for Part B, therefore, only Parts A and C results are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Primary Outcome: Overall Response Rate as Assessed by RECIST 1.1 Criteria
Time Frame: Up to end of study (up to 163 days)
Population: Data were not collected for the prespecified analysis of this outcome measure. No participants were enrolled for Part B.
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Complete and Partial Response Rate as Assessed by RECIST 1.1 Criteria
Time Frame: Up to end of study (up to 163 days)
Population: Data were not collected for the prespecified analysis of this outcome measure. No participants were enrolled for Part B.
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response
Time Frame: Up to end of study (up to 163 days)
Population: Data were not collected for the prespecified analysis of this outcome measure. No participants were enrolled for Part B.
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression-free Survival as Assessed by Per RECIST 1.1 Criteria
Time Frame: Up to end of study (up to 163 days)
Population: Data were not collected for the prespecified analysis of this outcome measure. No participants were enrolled for Part B.
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival as Assessed by Per RECIST 1.1 Criteria
Time Frame: Up to end of study (up to 163 days)
Population: Data was not collected for the prespecified analysis of this outcome measure. No participants were enrolled for Part B.
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pharmacokinetics: Maximum Observed Serum Concentration
Time Frame: Predose up to end of study (up to 163 days)
Population: Analysis was not performed as data were not collected for this outcome measure due to early study termination. No participants were enrolled for Part B.
Groups:
- XmAb18087 Monotherapy: Participants administered XmAb18087 Monotherapy.
Arm/Group | XmAb18087 Monotherapy
Number analyzed (Participants) | 0

8. Secondary Outcome: Immunogenicity: Number of Participants With Anti-XmAb18087 Antibodies
Time Frame: Up to end of study (up to 163 days)
Population: as for outcome 7
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) up to end of study (up to 163 days)
Arm/Group | Part A: XmAb18087 Monotherapy | Part C: XmAb18087 Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/2 | 2/2
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: XmAb18087 Monotherapy (N=2) | Part C: XmAb18087 Monotherapy (N=2)
Nausea (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: XmAb18087 Monotherapy (N=2) | Part C: XmAb18087 Monotherapy (N=2)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
gamma-glutamyltransferase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated by the sponsor and only 2 participants each were enrolled in Parts A and C. No participants were enrolled for Part B. Data were not collected for the prespecified analyses of efficacy, pharmacokinetics, and immunogenicity outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT04590781/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04590781/SAP_001.pdf